CLINICAL TRIAL: NCT00656370
Title: The INcreased Flow Utilizing Subcutaneously-Enabled Normal Saline and Lactated Ringer's (INFUSE-NSLR) Study: A Phase IV, Double-Blind, Randomized Study of Subcutaneous Hydration Enabled by Human Recombinant Hyaluronidase (Hylenex) in Volunteer Subjects
Brief Title: Study of Subcutaneous Hydration Enabled by Human Recombinant Hyaluronidase (Hylenex)
Acronym: INFUSE-NSLR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZ2-07-03
Record Dates: First submitted 2008-04-03; First posted 2008-04-11 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Hylenex; subcutaneous infusion; hyaluronidase; rHuPH20; recombinant human hyaluronidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NS Infusion Group (Experimental): Normal Saline (NS) and Hylenex
  Interventions: Drug: recombinant human hyaluronidase
- LR Infusion Group (Experimental): Lactated Ringer's (LR) and Hylenex
  Interventions: Drug: recombinant human hyaluronidase

INTERVENTIONS:
Drug: recombinant human hyaluronidase — 150 Units in 1mL
  Other Names: Hylenex

SUMMARY:
Randomized, double-blinded study that will evaluate the tolerability, safety, and flow rates of different solutions subcutaneously (SC) infused and preceded by human recombinant hyaluronidase (hylenex) 150 units.

In Stage 1, the comparison will be Normal Saline (NS) solution to Lactated Ringer's (LR) solution. Each subject will receive 500 milliliters (mL) of solution, consisting of NS in one thigh and LR in the other thigh. Immediately prior to the infusions, each thigh will have 150 units of hylenex.

In Stage 2, the comparison will be NS solution and buffered NS solution.

DETAILED DESCRIPTION:
This Phase IV, randomized, double-blinded study in volunteer subjects to evaluate the tolerability, safety, and flow rates of different solutions subcutaneously (SC) infused and preceded by human recombinant hyaluronidase (hylenex) 150 units. The study will be conducted in two sequential stages.

In Stage 1, the comparison will be NS solution to LR solution. Each subject will receive simultaneous SC infusions of 500 mL (from a 500 mL bag) of solution in each anterior thigh, consisting of NS in one thigh and LR in the other thigh. The thighs (left vs. right) to receive NS and LR will be randomized and double blinded. Immediately prior to the infusions, each thigh will have 150 units of hylenex simultaneously injected.

Tolerability will be assessed based on the subject's self-assessment of discomfort on a visual analog scale (VAS). Safety will be assessed by physical examination targeted at infusion sites, vital signs, and adverse events. The amount of fluid infused will be assessed by weighing the infusion bag, fluid and tubing at designated time points, and allowing the determination of flow rate.

Stage 2 will be conducted only if the observed Stage 1 VAS mean maximum pain score is at least 25 mm higher for one solution compared to the other. Stage 2 will evaluate the tolerability, safety, and flow rates of subcutaneously infused NS solution and buffered NS solution.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 60 years of age.
2. Intact normal skin without in the areas intended for infusion.
3. No fluid intake for 12 hours prior to the start of the study infusion.
4. Vital signs (Blood Pressure (BP), Heart Rate (HR), Respiratory Rate (RR)) within normal range.
5. Metabolic panel within normal range.
6. A negative urine or serum pregnancy test.
7. Signed, written Institutional Review Board (IRB)-approved informed consent.

Exclusion Criteria:

1. Lower extremity edema.
2. Lower extremity pathology that could interfere with study outcome.
3. Rales on lung auscultation.
4. History of cardiovascular disease.
5. Allergy to hyaluronidase.
6. Allergy to bee or vespid venom.
7. Pregnancy or breast-feeding woman.
8. Use of any investigational drug or device within 30 days of enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2008-01-30 (Actual); Study Completion 2008-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanthini Daniel, M.D., Principal Investigator — Jasper Clinic, Inc.
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject entered screening on 19 DEC 2007 and the last subject entered screening on 23 JAN 2008. A total of 25 subjects were assessed for eligibility and signed an Informed Consent Form.
Pre-assignment Details: Seven subjects were excluded during screening: 6 did not meet inclusion criteria and 1 withdrew consent. An additional 3 subjects were screened as alternates, but were not enrolled. 15 subjects were randomized and completed stage 1.
Groups:
- NS, LR: In Stage 1, the comparison will be NS solution to LR solution. Each subject will receive simultaneous SC infusions of 500 mL (from a 500 mL bag) of solution in each anterior thigh, consisting of NS in one thigh and LR in the other thigh. The thighs (left vs. right) to receive NS and LR will be randomized and double blinded. Immediately prior to the infusions, each thigh will have 150 units of hylenex simultaneously injected.
Period: Overall Study
Arm/Group | NS, LR
Started | 25 (25 subjects were assessed for eligibility and signed an Informed Consent Form.)
Completed | 15 (15 subjects were randomized and completed stage 1 (received both NS and LR).)
Not Completed | 10
Not completed — Screen Failures | 7
Not completed — Alternates | 3

BASELINE CHARACTERISTICS:
Arm/Group | NS, LR
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: The Participant's Assessment of Discomfort at the Infusion Site on a Visual Analog Scale (VAS)
Description: Participant's self-assessment of discomfort at the infusion site by means of a validated VAS with a range of 0 millimeters (mm) (no discomfort) to 100 mm (worst possible discomfort), for the comparison of subcutaneous (SC) infusion of normal saline (NS) versus Lactated Ringer's (LR), each following an SC slow-push injection of 150 Units (U) Hylenex.
Time Frame: Approximate times which ranged from zero minutes at baseline to maximal post-infusion of 240 minutes on Day 1
Population: 15 subjects were randomized and completed stage 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | NS Infusion Group | LR Infusion Group
Number analyzed (Participants) | 15 | 15
mm | 20.0 (19.4) | 9.4 (18.3)

2. Secondary Outcome: Number of Participants Assessed for Safety Measures
Description: Safety outcome measures included adverse events (AEs), physical examinations (targeted physical examination included lung auscultation for rales, checking for edema, evaluation of infusion sites, positives on a review of systems, and follow-up of findings from previous physical examinations), and vital signs (systolic blood pressure, diastolic blood pressure, heart rate, and respiration rate).
Time Frame: Baseline, Mid-Infusion Right and Left, Post-Infusion Right and Left, Discharge Right and Left (up to approximately 8 days)
Population: 15 participants were randomized and completed stage 1
Measure: Number; unit: participants
Arm/Group | NS, LR
Number analyzed (Participants) | 15
participants | 15

3. Secondary Outcome: Average Infusion Flow Rate (Milliliters Per Hour [mL/hr]) Derived From the Time to Infuse up to 500 mL of Solution
Description: The infusion flow rate (mL/h) was derived from the time to subcutaneously (SC) infuse up to 500 mL of NS or LR solution (following SC injection of 150 Units hylenex) by measuring the change in weight of the infusion bag, fluid, and tubing.
Time Frame: During infusion on Day 1
Population: 15 participants were randomized and completed stage 1
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | NS Infusion Group | LR Infusion Group
Number analyzed (Participants) | 15 | 15
mL/hr | 384.1 (118.1) | 395.8 (132.8)
Statistical Analysis 1: Comparison: NS Infusion Group vs LR Infusion Group; Test type: Superiority; p = 0.93, Wilcoxon signed rank test

4. Secondary Outcome: Percent Change From Baseline Thigh Circumference to Maximum Post-Baseline Thigh Circumference at Infusion Sites
Description: Thigh circumference was measured in centimeters at 7 time points before, during, and after subcutaneous infusion of 500 mL NS or LR solution.
Time Frame: Before the infusion, during the infusion, after the infusion, and discharge (Day 1)
Population: 15 participants were randomized and completed stage 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NS Infusion Group | LR Infusion Group
Number analyzed (Participants) | 15 | 15
percent change | 5.2 (1.6) | 5.3 (1.5)
Statistical Analysis 1: Comparison: NS Infusion Group vs LR Infusion Group; Test type: Superiority; p = 0.67, Wilcoxon signed rank test

5. Secondary Outcome: Time From the Beginning of Infusion Until the Thigh Circumference Returns to Within 5% of Baseline Circumference
Description: Thigh circumference was measured at the level of the angiocatheter with a flexible measuring tape prior to infusion initiation (Baseline), at the midpoint for each infusion, and at the end of each infusion.
Time Frame: Before the infusion (Baseline) until discharge (Day 1)
Population: 15 participants were randomized and completed stage 1. Only those participants who experienced a 5% or greater increase in thigh circumference for both infusions were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NS Infusion Group | LR Infusion Group
Number analyzed (Participants) | 4 | 4
minutes | 147.3 (35.6) | 123.5 (9.7)

6. Secondary Outcome: Number of Participant's With the Indicated Global Preference for Infusion (Left Versus Right Thigh)
Description: Participants blinded to the type of infusion were asked to state their preference for the left or right infusion following all infusion day (Day 1) activities and assessments. The preference for the left or right infusion indicated which infusion was preferred: NS or LR.
Time Frame: End of infusion (Day 1)
Population: 15 participants were randomized and completed stage 1
Measure: Count of Participants; unit: Participants
Arm/Group | NS Infusion Group | LR Infusion Group
Number analyzed (Participants) | 15 | 15
Participants | 0 | 15

ADVERSE EVENTS:
Arm/Group | NS, LR
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NS, LR (N=15)
Injection site pain (General disorders) | 11 (16)
Injection site erythema (General disorders) | 7 (9)
Injection site irritation (General disorders) | 4 (7)
Injection site pruritus (General disorders) | 2 (3)
Injection site bruising (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless prior written permission from the Sponsor (Halozyme) is obtained.